CLINICAL TRIAL: NCT03070171
Title: Bioequivalence of Tablet Formulation of Dabigatran Etexilate Compared to Commercial Capsule Formulation Following Oral Administration in Healthy Male Subjects (an Open-label, Randomised, Single-dose, Replicate Design in a Two-treatment, Four-period, Two-sequence Crossover Study)
Brief Title: Bioequivalence of Tablet Formulation of Dabigatran Etexilate Compared to Commercial Capsule Formulation Following Oral Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160-0271
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dabigatran Etexilate Capsule (Experimental)
  Interventions: Drug: dabigatran etexilate
- Dabigatran Etexilate Tablet (Experimental)
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — single dose
  Other Names: PRADAXA

SUMMARY:
The primary objective of this trial is to establish the bioequivalence of tablet formulation of dabigatran etexilate compared to commercial capsule formulation following oral administration under fasted condition.

The secondary objective is the evaluation and comparison of several pharmacokinetic parameters between the treatments.

ELIGIBILITY:
Inclusion Criteria:

Subjects will only be included into the trial, if they meet the following criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age ≥20 and ≤40 years old at informed consent
* BMI ≥18 and ≤25 kg/m2 at screening
* Signed and dated written informed consent prior to admission to the trial in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

Subjects will not be allowed to participate if any of the following general criteria apply:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR)or electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm at screening. Based on the clinical judge by the investigator, repeated measurements are allowed.
* Any laboratory value outside the reference range before randomisation that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease considered as clinically relevant by the investigator
* Any relevant bleeding history considered by the investigator
* Any history or evidence of blood dyscrasia, haemorrhagic diathesis, severe thrombocytopenia, cerebrovascular haemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with haemorrhagic tendencies
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Planned surgeries within four weeks following the end-of trial examination
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl.Qc/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking in-house confinement at the trial site
* Alcohol abuse (consumption of more than 30 g per day: e.g., 750 mL of beer, 1.5 gous [equivalent to 270 mL] of Sake)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with trial requirements, or has a condition that would not allow safe participation in the trial

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

REFERENCES:
- [Derived] Harada A, Ikushima I, Haranaka M, Yanagihara A, Nakayama D. Bioequivalence of a Newly Developed Dabigatran Etexilate Tablet Versus the Commercial Capsule and Impact of Rabeprazole-Induced Elevated Gastric pH on Exposure in Healthy Subjects. Am J Cardiovasc Drugs. 2020 Jun;20(3):249-258. doi: 10.1007/s40256-019-00377-x. PMID 31667735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomised, single-dose, open-label, replicate design in a two-treatments, four-period, two-sequence crossover design (T:Dabigatran etexilate tablet formulation 110 mg and R: Dabigatran etexilate capsule formulation 110 mg)
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Groups:
- T-R-R-T: Subjects were treated with single oral dose, started in period 1 with 110 milligram (mg) Dabigatran etexilate tablet with 200 milliliter (mL) of water after an overnight fast of at least 10 hour (h), followed in period 2 and period 3 by 110 mg Dabigatran etexilate capsule with 200 mL of water after an overnight fast of at least 10 h, and in period 4 by 110 mg Dabigatran etexilate tablet with 200 mL of water after an overnight fast of at least 10 h. Treatment periods were separated by a wash-out phase of at least 4 days.
- R-T-T-R: Subjects were treated with single oral dose, started in period 1 with 110 mg Dabigatran etexilate capsule with 200 mL of water after an overnight fast of at least 10 h, followed in period 2 and period 3 by 110 mg Dabigatran etexilate tablet with 200 mL of water after an overnight fast of at least 10 h, and in period 4 by 110 mg Dabigatran etexilate capsule with 200 mL of water after an overnight fast of at least 10 h. Treatment periods were separated by a wash-out phase of at least 4 days.
Period: Treatment Period 1 + Washout
Arm/Group | T-R-R-T | R-T-T-R
Started | 80 | 80
Completed | 80 | 80
Not Completed | 0 | 0
Period: Treatment Period 2 + Washout
Arm/Group | T-R-R-T | R-T-T-R
Started | 80 | 80
Completed | 80 | 79
Not Completed | 0 | 1
Not completed — Other Adverse Event | 0 | 1
Period: Treatment Period 3 + Washout
Arm/Group | T-R-R-T | R-T-T-R
Started | 80 | 79
Completed | 80 | 79
Not Completed | 0 | 0
Period: Treatment Period 4 + Washout
Arm/Group | T-R-R-T | R-T-T-R
Started | 80 | 79
Completed | 80 | 78
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects from the Randomised Set (RS) who were dispensed study medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | T-R-R-T | R-T-T-R | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: TS
  Years | 27.2 (4.2) | 27.3 (4.2) | 27.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 0 | 0 | 0
    Male | 80 | 80 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 80 | 80 | 160
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 80 | 80 | 160
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz of Free Dabigatran
Description: Area under the concentration-time curve of free dabigatran in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz). Geometric Mean (gMean) is actually Adjusted gMean & Geometric Coefficient of Variation (gCV) is actually Intra individual gCV (%gCV).
  PK exclusion criteria: 1) The subject experienced emesis at or before 2 times median Time from (last) dosing to the maximum measured concentration of the analyte in plasma (tmax). Median tmax was to be taken either from the median tmax for reference product or test product, depending on whether the subject had experienced emesis after taken the test or reference product. Median tmax was to be determined excluding the subjects experiencing emesis. 2) Time deviations 3) Use of restricted medications 4) A pre-dose concentration was >5% of the Cmax value of that subject.
Time Frame: 1:00h before drug administration and 0:30h, 1:00h, 1:30h, 2:00h, 3:00h, 4:00h, 6:00h, 8:00h, 12:00h, 24:00h, 36:00h and 48:00h after drug administration.
Population: Pharmacokinetic set (PKS): All subjects from Treated Set (TS) who provided at least 1 observation for at least 1 primary endpoint that was not excluded as per PK exclusion criteria (defined in the description).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng･h/mL)
Groups:
- Dabigatran Etexilate Tablet (T): Patients were administered single oral dose of 110 mg Dabigatran etexilate tablet with 200 mL of water after an overnight fast of at least 10 h
- Dabigatran Etexilate Capsule (R): Patients were administered single oral dose of110 mg Dabigatran etexilate capsule with 200 mL of water after an overnight fast of at least 10 h
Arm/Group | Dabigatran Etexilate Tablet (T) | Dabigatran Etexilate Capsule (R)
Number analyzed (Participants) | 159 | 160
Nanogram*hour/milliliter (ng･h/mL) | 725.03686 (57.00406) | 668.42714 (52.33393)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet (T) vs Dabigatran Etexilate Capsule (R); The statistical model was an analysis of variance (ANOVA) on the logarithmic scale including effects for 'sequence', 'subjects nested within sequences', 'period' and 'treatment'; Test type: Equivalence — Bioequivalence was established by ensuring that the T/R ratio of AUC0-tz of free dabigatran was within the pre-specified acceptance range (80%-125%); ANOVA; T/R Ratio = 108.46909, 90% CI 2-sided [101.44605 to 115.97833] — Confidence intervals were calculated based on the residual error from ANOVA. Ratio calculated as Dabigatran Etexilate Tablet (T) divided by Dabigatran Etexilate capsule (R)

2. Primary Outcome: Cmax of Free Dabigatran
Description: Maximum plasma concentration of free dabigatran (Cmax). Geometric Mean is actually Adjusted geometric mean and Geometric Coefficient of Variation (gCV) is actually Intra individual gCV.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Dabigatran Etexilate Tablet (T) | Dabigatran Etexilate Capsule (R)
Number analyzed (Participants) | 159 | 160
Nanogram/milliliter (ng/mL) | 86.26026 (56.43338) | 79.16785 (55.20456)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet (T) vs Dabigatran Etexilate Capsule (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Bioequivalence was established by ensuring that the T/R ratio of Cmax of free dabigatran was within the pre-specified acceptance range (80%-125%); ANOVA; T/R Ratio = 108.9587, 90% CI 2-sided [101.78627 to 116.63654] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: AUC0-tz of Total Dabigatran
Description: Area under the concentration-time curve of total dabigatran in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz ).
  Geometric Mean is actually Adjusted geometric mean and Geometric Coefficient of Variation (gCV) is actually Intra individual gCV.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | Dabigatran Etexilate Tablet (T) | Dabigatran Etexilate Capsule (R)
Number analyzed (Participants) | 159 | 160
ng•h/mL | 847.26720 (57.32236) | 787.31279 (52.53129)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet (T) vs Dabigatran Etexilate Capsule (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; ANOVA; T/R Ratio = 107.61507, 90% CI 2-sided [100.61938 to 115.09714] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax of Total Dabigatran
Description: Maximum plasma concentration of total dabigatran (Cmax). Geometric Mean is actually Adjusted geometric mean and Geometric Coefficient of Variation (gCV) is actually Intra individual gCV.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate Tablet (T) | Dabigatran Etexilate Capsule (R)
Number analyzed (Participants) | 159 | 160
ng/mL | 99.81133 (58.31846) | 93.54769 (56.54651)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet (T) vs Dabigatran Etexilate Capsule (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Bioequivalence was established by ensuring that the T/R ratio of Cmax of total dabigatran was within the pre-specified acceptance range (80%-125%); ANOVA; T/R Ratio = 106.69566, 90% CI 2-sided [99.50139 to 114.41010] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: AUC0-∞ of Total Dabigatran
Description: Area under the concentration-time curve of total dabigatran in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Geometric Mean is actually Adjusted geometric mean and Geometric Coefficient of Variation (gCV) is actually Intra individual gCV.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | Dabigatran Etexilate Tablet (T) | Dabigatran Etexilate Capsule (R)
Number analyzed (Participants) | 159 | 160
ng•h/mL | 877.70198 (52.04260) | 813.94379 (49.99079)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet (T) vs Dabigatran Etexilate Capsule (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Bioequivalence was established by ensuring that the T/R ratio of AUC0-∞ of total dabigatran was within the pre-specified acceptance range (80%-125%); ANOVA; T/R Ratio = 107.83324, 90% CI 2-sided [101.25584 to 114.83790] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: AUC0-∞ of Free Dabigatran
Description: Area under the concentration-time curve of free dabigatran in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Geometric Mean is actually Adjusted geometric mean and Geometric Coefficient of Variation (gCV) is actually Intra individual gCV.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•h/mL
Arm/Group | Dabigatran Etexilate Tablet (T) | Dabigatran Etexilate Capsule (R)
Number analyzed (Participants) | 159 | 160
ng•h/mL | 753.13668 (51.62318) | 694.57320 (49.42941)
Statistical Analysis 1: Comparison: Dabigatran Etexilate Tablet (T) vs Dabigatran Etexilate Capsule (R); [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Bioequivalence was established by ensuring that the T/R ratio of AUC0-∞ of free dabigatran was within the pre-specified acceptance range (80%-125%); ANOVA; T/R Ratio = 108.43158, 90% CI 2-sided [101.87254 to 115.41292] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration until 3 day after the last drug administration, ie upto 7 days
Arm/Group | Dabigatran Etexilate Tablet (T) | Dabigatran Etexilate Capsule (R)
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/160
Other Adverse Events (participants affected / at risk) | 0/159 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03070171/SAP_000.pdf
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03070171/Prot_001.pdf